CLINICAL TRIAL: NCT06302062
Title: An Open,Single-center,Phase I Clinical Study of Tumor-associated Lymph Node T Cell Therapy for Advanced Solid Tumors
Brief Title: Phase I Clinical Study of Tumor-associated Lymph Node T Cell Therapy for Advanced Solid Tumors
Acronym: TAL-T
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou FineImmune Biotechnology Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIT003-IIT
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumor; Tumor Associated Lymph Node T Cell; Immunotherapy
Keywords: TAL-T; cell therapy; Tumor Associated Lymph node T cell; Safety; Adverse Drug Event; Efficacy; Immunotherapy; Serplulimab Injection
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Cyclophosphamide; Interleukin-2; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Three patients were planned to be enrolled, and each subject received one to two cell transfusions.
  Interventions: Drug: Tumor Associated Lymph node T cell; Drug: cyclophosphamide; Drug: IL-2
- Cohort B (Experimental): 14 to 20 patients were enrolled, and each subject received one to two cell transfusions. In this group, Tumor Associated Lymph node T cells were combined with Serplulimab Injection.
  Interventions: Drug: Tumor Associated Lymph node T cell; Drug: cyclophosphamide; Drug: IL-2; Drug: Serplulimab Injection

INTERVENTIONS:
Drug: Tumor Associated Lymph node T cell — At least one lymph sample is resected from each participant, then it is separated and cultured ex vivo to expand the population of Tumor Associated Lymph node T cells (FIT003 TAL-T). After lymphodepletion, patients are infused with FIT003 TAL-T.
  Other Names: TAL-T cells; TAL-T
Drug: cyclophosphamide — A one-day intravenous injection of cyclophosphamide was administered two days prior to the initial cell transfusion.
Drug: IL-2 — The IL-2 treatment will be continued for 5 days.
  Other Names: Cellular interleukin 2; interleukin-2
Drug: Serplulimab Injection — In group B, Serplulimab Injection was injected before and after cell transfusion. If two cell transfusions were performed,Serplulimab Injection were given again .
  Other Names: PD1 monoclonal antibody; PD1
  Arms: Cohort B

SUMMARY:
A total of 17 to 23 participants are anticipated to be enrolled in the Phase I clinical trial, which is further divided into two distinct parts: one part involves single-agent cell therapy, while the other entails a combination of cell therapy and Serplulimab Injection.

To be more precise, the study aims to include patients who have been diagnosed with metastatic or locally advanced refractory/recurrent malignant solid tumors and have shown resistance to standard therapeutic interventions. These tumor types may encompass head and neck cancer, ovarian cancer, lung cancer, melanoma, and others.

DETAILED DESCRIPTION:
This is an open, single-center Phase I clinical trial designed to assess the safety, tolerability, efficacy, and feasibility of tumor-associated lymph node T cells (TAL-T) for treating metastatic solid tumors. The study consists of three distinct phases: screening, administration of treatment, and follow-up evaluation. In this investigation, TAL-T cells will be cultured after being separated in a laboratory setting. Participants will receive 1-2 infusions of TAL-T cells.

ELIGIBILITY:
Before conducting tumor-associated lymph node sampling, it is necessary to verify that subjects meet the inclusion criteria marked with an asterisk (*). These criteria include:

1. * being between the ages of 18 and 75;
2. having metastatic or locally advanced refractory/recurrent malignant solid tumors that have failed standard therapy or have failed to tolerate standard treatment;
3. having at least one measurable target lesion;
4. * voluntarily participating and signing an informed consent form;
5. * having at least one resectable tumor-associated lymph node from which T cells can be successfully isolated;
6. * having an ECOG score of 0-1;
7. * having an expected survival of more than 6 months;
8. * female subjects with fertility potential must have a negative pregnancy test, and all men and women with fertility potential must consent to using medically effective contraception during the study period and for 12 months after the last dose of the study medication;
9. * being willing to regularly come to the hospital for treatment, testing, evaluation, and management as required during the entire study period.

Before sampling tumor-associated lymph nodes, it is important to confirm that the subject does not meet any of the exclusion criteria marked with an asterisk (*). These criteria include：

1. * Experiencing moderate to severe infection or at risk of opportunistic infection;
2. * Present with active autoimmune disease (other than vitiligo or childhood asthma/allergies that have healed);
3. * Uncontrolled concomitant disease, including but not limited to symptomatic congestive heart failure, unstable angina pectoris, arrhythmias (excluding stable atrial fibrillation), and significant carotid stenosis.
4. * Acute systemic infections, coagulation disorders or other serious cardiopulmonary diseases;
5. Patients who have used large amounts of glucocorticoids or other immunosuppressants within 4 weeks;
6. * A history of severe hypersensitivity to any of the drugs used in this study;
7. Known uncontrolled central nervous system (CNS) metastases and/or cancerous meningitis;
8. * Pregnant and lactating women, as well as women and men who were unable to cooperate with contraception during the study period;
9. Previous anti-tumor therapy: within four weeks of radiotherapy, chemotherapy, one week after TKI inhibitor treatment, four weeks of investigational therapy or four half-lives, whichever is shorter;
10. * Enroll in another clinical study at the same time, unless it is an observational, non-interventional clinical study or the follow-up period of an interventional study;
11. * Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
12. * Known history of interstitial lung disease. Exclude subjects with high suspicion of interstitial pneumonia; Or may interfere with the detection or management of suspected drug-related pulmonary toxicity; Or other moderate to severe lung diseases that seriously affect lung function;
13. * Known history of primary immunodeficiency virus infection or positive HIV test;
14. * Patients with chronic hepatitis B or HBV carriers of chronic hepatitis B virus (HBV), or patients with active hepatitis C should be excluded;
15. * Any of the following cardiovascular diseases

    1. have evidence of acute or persistent episodes of myocardial ischemia;
    2. symptomatic pulmonary embolism is present;
    3. acute myocardial infarction occurred within 6 months prior to the initial study treatment;
    4. symptomatic congestive heart failure (grade 3 or 4 according to the New York Heart Association Functional Scale) occurred within 6 months prior to the first study treatment;
    5. Occurrence of grade 2 or more ventricular arrhythmias within 6 months prior to the first study treatment;
    6. cerebrovascular accident or transient ischemic stroke occurred within 6 months prior to the first study treatment
16. * Subjects with pleural effusion, pericardial effusion, or ascites that, in the investigator's judgment, cannot be stably controlled by repeated drainage or other methods;
17. Have received a live vaccine within 30 days prior to the first dose or plan to receive a live vaccine during the study period;
18. * Disease known to produce severe hypersensitivity to other monoclonal antibodies;
19. Any condition that the investigator believes may result in a risk of acceptance of the study drug treatment or interfere with the evaluation of the study drug or the safety of the subjects or the interpretation of the study results;
20. * With a second primary tumor (within 5 years).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DLT | At least 58 days
  The dosage of TAL-T was determined to limit toxicity
MDT | At least 58 days
  Determine the maximum tolerated dose of TAL-T
Number of participants with treatment-related adverse events as assessed by CTCAE V4.03 | At least 60 days
  Keep record the adverse eventd experienced by subjects in 30 days after the last infusion

SECONDARY OUTCOMES:
ORR | one yaer
  The proportion of subjects receiving a confirmed optimal response of PR or above which was evaluation according to RECIST or iRECIST principles.
PFS | two years
  The time between the subject receiving treatment and the onset of PD or death from any cause, whichever occurs first. If the subject had no events (PD or death), the last response assessment day was the cut-off time for PFS.
life quality score | At least 70 days
  ECOG 0-1

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Gaungdong, China